CLINICAL TRIAL: NCT06008314
Title: Development of "SMART on FHIR (Fast Healthcare Interoperability Resources)" Interoperable Clinical Decision Support (CDS) for Emergency Department (ED) Patients With Pneumonia & Pilot Deployment Into Novel Epic Electronic Health Record (EHR) Environments
Brief Title: Pilot Deployment of ePNa Into Epic EHR
Acronym: ePNa-Epic
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nathan Dean (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency); Vanderbilt University (Other); Stanford University (Other)
Responsible Party: Sponsor-Investigator, Nathan Dean, Professor, Pulmonary and Critical Care Medicine, Intermountain Health Care, Inc.
Organization: Intermountain Health Care, Inc. (Other)
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 1052404
Record Dates: First submitted 2023-08-04; First posted 2023-08-23 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Pneumonia
Keywords: Decision Support
MeSH Terms: conditions — Pneumonia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Implementation at Vanderbilt University Medical Center (VUMC) & Vanderbilt Wilson County Hospital (Experimental): ePNa (the decision support tool) will be implemented at 2 EDs that are part of the Vanderbilt Health system.
  Interventions: Other: ePNa

INTERVENTIONS:
Other: ePNa — Real-time, automated clinical decision support tool for pneumonia (called "ePNa")

SUMMARY:
Intermountain Health has developed a electronic decision support tool to help doctors provide the best care for pneumonia. The purpose of this study is to enhance the existing tool (called ePneumonia (electronic Pneumonia) or ePNa) so that it can be used at other institutions, and to test deployment of the tool at another institution's hospitals.

DETAILED DESCRIPTION:
This study as funded by the AHRQ (Agency for Healthcare Research and Quality) involves making the current ePNa system a "SMART on FHIR" compatible application that will enable the same core software and processes to work across the Cerner and Epic electronic health record platforms. The investigators will then engage with emergency department providers and patients to improve user centered design, considering clinician preferences and feedback for use as well as patient needs for information. Finally, the investigators will evaluate the feasibility and acceptability via a pilot implementation trial of the interoperable ePNa platform at two Vanderbilt affiliated hospitals.

ELIGIBILITY:
Inclusion Criteria:

For the baseline database and assessment of clinical outcomes, all data will be pulled from the Epic Clarity data warehouse.

* 2500 patients that presented to the Vanderbilt and Wilson county EDs who are >= 18 years old will be identified by ICD-10 codes for pneumonia or acute respiratory failure or sepsis with secondary pneumonia codes for the baseline database.
* An additional 2500 patients that presented to the Vanderbilt and Wilson county EDs who are >= 18 years old will be identified by having had conventional PA (posteroanterior) and lateral or portable CXRs (chest X-rays), independent of ICD-10 codes.
* During the one year pilot trial, patients seen in the 2 EDs, who are >= 18 years old will be identified by ICD(International Classification of Diseases)-10 codes for pneumonia or acute respiratory failure or sepsis with secondary pneumonia codes (estimated to comprise 1800 patients).

Exclusion Criteria:

For all above patients:

1. Patients seen with a history of recent trauma.
2. Subsequent episodes of pneumonia from the same patient within the study period.
3. Patients directly admitted to hospice/comfort care.
4. Patients admitted to a non-study hospital for further care.
5. Patients transferred from outside hospitals.

For the groups selected by ICD-10 pneumonia codes, an additional exclusion is:

• Patients without radiographic evidence of pneumonia or with clear radiographic evidence for an alternative diagnosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6917 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
14-day hospital-free days | 14 days after initial presentation to the emergency department
  14-day hospital-free days (a metric which captures outpatient disposition from the emergency department, secondary hospital admission, and length of stay)

SECONDARY OUTCOMES:
30-day all-cause mortality | At 30 days after initial ED presentation
ED length of stay (hours) | At ED discharge
ICU length of stay (days) | At ICU discharge
Number of patients admitted to floor who are subsequently transferred to ICU within 72 hours | At 72 hours after inpatient admission
Time from ED presentation to first antibiotic dose (minutes) | At time of first antibiotic dose

CONTACTS AND LOCATIONS:
Overall Officials: Nathan Dean, MD, Principal Investigator — Intermountain Health

IPD SHARING:
Plan to Share IPD: No